CLINICAL TRIAL: NCT05030506
Title: An Open-Label, Phase 1 Study of MK-6482 as Monotherapy and in Combination With Lenvatinib (MK-7902) With or Without Pembrolizumab (MK-3475) in China Participants With Advanced Renal Cell Carcinoma
Brief Title: A Study of Belzutifan (MK-6482) as Monotherapy and in Combination With Lenvatinib (E7080/MK-7902) With or Without Pembrolizumab (MK-3475) in China Participants With Advanced Renal Cell Carcinoma (MK-6482-010)
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6482-010; MK-6482-010 (Other: MSD)
Record Dates: First submitted 2021-08-30; First posted 2021-09-01 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Renal Cell Carcinoma
Keywords: Belzutifan; Pembrolizumab; Programmed Cell Death-1 (PD1); Hypoxia inducible factor 2 alpha (HIF-2 alpha); Hypoxia inducible factor 2α (HIF-2α); Renal Cell Carcinoma (RCC); Kidney Cancer; MK-6482; MK6482; PT-2977; PT2977; MK-3475 KEYTRUDA®; MK-7902; E7080; LENVIMA®
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms | interventions — belzutifan; pembrolizumab; lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Belzutifan + Lenvatinib (Experimental): Participants will receive a daily oral dose of 120 mg of belzutifan monotherapy for 3 weeks, followed by a combination of a daily oral dose of 120 mg of belzutifan with a daily oral dose of 20 mg of lenvatinib until progressive disease or discontinuation.
  Interventions: Drug: Belzutifan; Drug: Lenvatinib
- Belzutifan + Lenvatinib + Pembrolizumab (Experimental): Participants will receive an intravenous dose of 400 mg of pembrolizumab once every six weeks for up to 18 infusions (up to 2 years) in combination with a daily oral dose of 120 mg of belzutifan and a daily oral dose of 20 mg of lenvatinib until progressive disease or discontinuation.
  Interventions: Drug: Belzutifan; Biological: Pembrolizumab; Drug: Lenvatinib

INTERVENTIONS:
Drug: Belzutifan — 40 mg tablet administered orally at a dose of 120 mg
  Other Names: MK-6482; PT2977
Biological: Pembrolizumab — 25 mg/mL solution for Infusion in a single-dose vial administered intravenously at a dose of 400 mg
  Other Names: MK-3475 KEYTRUDA®
  Arms: Belzutifan + Lenvatinib + Pembrolizumab
Drug: Lenvatinib — 10 mg capsule administered orally at a dose of 20 mg
  Other Names: MK-7902; E7080; LENVIMA®

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetic and pharmacodynamic profiles, and preliminary efficacy of belzutifan as monotherapy followed by belzutifan+lenvatinib combination therapy, as well as belzutifan combined with lenvatinib and pembrolizumab in China participants with advanced renal cell carcinoma.

ELIGIBILITY:
Inclusion Criteria

* Has a histologically confirmed diagnosis of unresectable, locally advanced or metastatic clear cell renal cell carcinoma (RCC).
* Has measurable disease per RECIST 1.1.
* Has adequate organ function.
* Has adequately controlled blood pressure (BP).
* If participants received major surgery or radiation therapy of >30 Gy, they must have recovered from the toxicity and/or complications from the intervention.
* Has resolution of the toxic effect(s) of the most recent prior therapy.
* Participants receiving bone resorptive therapy must have therapy initiated at least 2 weeks prior to allocation.
* Is Chinese descent, defined as both biological parents and all biological grandparents are of Chinese descent.

Male Participants:

- Must be willing to use an adequate method of contraception.

Female Participants:

- Must be a woman of non-childbearing potential (WONCBP) or have a negative urine or serum pregnancy test and must be willing to use an adequate method of contraception.

For Belzutifan + Lenvatinib treatment:

* Has progressed on or after having received systemic treatment for locally advanced or metastatic RCC.
* Has no more than 3 prior systemic regimens for locally advanced or metastatic RCC.

For Belzutifan + Lenvatinib + Pembrolizumab treatment:

- Has received no prior systemic therapy for advanced RCC.

Exclusion Criteria

* Is a woman of childbearing potential (WOCBP) who has a positive urine pregnancy test within 24 hours prior to first dose of study intervention.
* Has any of the following: A pulse oximeter reading <92%, or requires intermittent supplemental oxygen, or requires chronic supplemental oxygen.
* Has a known additional malignancy that is progressing or has required active treatment within the past 3 years.
* Has known central nervous system (CNS) metastases and/or carcinomatous meningitis.
* Has clinically significant cardiac disease.
* Has symptomatic pleural effusion.
* Has a history of inflammatory bowel disease.
* Has preexisting ≥Grade 3 gastrointestinal or non-gastrointestinal fistula.
* Has clinically significant hematuria, hematemesis or hemoptysis of red blood, or other history of significant bleeding within 3 months before administration of the first dose of study intervention.
* Has other clinically significant disorders such as: A serious active non-healing wound/ulcer/bone fracture, requirement for hemodialysis or peritoneal dialysis or a history of allogenic tissue/solid organ transplantation.
* Received colony-stimulating factors, granulocyte macrophage colony-stimulating factor (GMCSF) or recombinant EPO within 28 days prior to the first dose of study intervention.
* Has a known psychiatric or substance abuse disorder that would interfere with cooperation with the requirements of the study.
* Is unable to swallow orally administered medication or has a gastrointestinal disorder affecting absorption.
* Has received prior treatment with belzutifan.
* Has received prior treatment with lenvatinib.
* Has received any type of systemic anticancer antibody (including investigational antibody) ≤28 days prior to allocation.
* Has received / will be receiving any traditional Chinese medicines.
* Has received prior radiotherapy within 2 weeks prior to first dose of study intervention. Participants must have recovered from all radiation-related toxicities and not require corticosteroids.
* Is receiving concomitant treatment, in therapeutic doses, with anticoagulants.
* Is receiving chronic systemic steroids therapy (at doses >10 mg daily of prednisone or equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study intervention.
* Is currently participating in a study of an investigational agent or is currently using an investigational device.
* Has an active infection requiring systemic therapy.
* Has a known history of Human Immunodeficiency Virus (HIV) infection.
* Has a known history of Hepatitis B or known active Hepatitis C virus infection.
* Has a known history of active tuberculosis.
* Has radiographic evidence of intratumoral cavitation, encasement or invasion of a major blood vessel.
* Has known hypersensitivity or allergy to the active pharmaceutical ingredient or any component of the study intervention (belzutifan or lenvatinib) formulations.
* Has had major surgery within 4 weeks prior to first dose of study intervention.

For Belzutifan + Lenvatinib + Pembrolizumab treatment:

* Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
* Has a history of hypersensitivity reaction to the active pharmaceutical ingredient or any component of pembrolizumab or monoclonal antibody (mAb).
* Has an active autoimmune disease that has required systemic treatment in the past 2 years.
* Has received a live vaccine within 30 days prior to the first dose of study intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2021-10-13 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants who experienced dose-limiting toxicities (DLTs) | Up to approximately 21 days
  A DLT is defined as an event with toxicity including the type, severity, time of onset, time of resolution, and the probable association with study treatment that are not due to pre-existing conditions as defined by the Common Terminology Criteria for Adverse Events Version 5.0 (CTCAE 5.0). Number of participants who experience a DLT per CTCAE 5.0 will be reported.
Number of participants who experienced an adverse event (AE) | Up to approximately 68 months
  An AE is any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening of a preexisting condition that is temporally associated with the use of the Sponsor's product, is also an AE. The number of participants who experience an AE in the study will be reported.
Number of participants who discontinued study treatment due to an AE | Up to approximately 68 months
  An AE is any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening of a preexisting condition that is temporally associated with the use of the Sponsor's product, is also an AE. The number of participants who discontinued from the study treatment due to an AE will be reported.
Area under the concentration-time curve from 0-24 hours (AUC0-24) of belzutifan after single dose (Cohort 1) | Pre-dose, and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours postdose
  AUC is a measure of plasma drug concentration and time and is estimated as the area under the plot of plasma concentration against time after drug administration. Blood samples collected pre dose and at multiple timepoints post dose will be used to determine AUC0-24 of belzutifan.
Maximum concentration (Cmax) of belzutifan after single dose (Cohort 1) | Pre-dose, and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours postdose
  Cmax is the maximum concentration of the drug observed in plasma. Blood samples collected pre dose and at multiple timepoints post dose will be used to determine Cmax of belzutifan.
Time at maximum concentration (Tmax) of belzutifan after single dose (Cohort 1) | Pre-dose, and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours postdose
  Tmax is the amount of time that a drug is present at the maximum concentration is observed in plasma. Blood samples collected pre dose and at multiple timepoints post dose will be used to determine the Tmax of belzutifan.
Steady state area under the concentration-time curve from 0-24 hours (AUC0-24,ss) of belzutifan after multiple doses (Cohort 1) | Pre-dose, and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours postdose
  AUC0-24,ss is a measure of plasma drug concentration and time and is estimated as the area under the plot of plasma concentration against time after drug administration. Blood samples collected pre dose and at multiple timepoints post dose will be used to determine AUC0-24,ss of belzutifan.
Steady state maximum concentration (Cmax,ss) of belzutifan after multiple doses (Cohort 1) | Pre-dose, and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours postdose
  Cmax,ss is the maximum concentration of the drug observed in plasma. Blood samples collected pre dose and at multiple timepoints post dose will be used to determine Cmax,ss of belzutifan.
Time at maximum concentration (Tmax) of belzutifan after multiple doses (Cohort 1) | Pre-dose, and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours postdose
  Tmax is the amount of time that a drug is present at the maximum concentration is observed in plasma. Blood samples collected pre dose and at multiple timepoints post dose will be used to determine the Tmax of belzutifan.
Apparent t½ of belzutifan after multiple doses (Cohort 1) | Pre-dose, and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours postdose.
  T1/2 is a measure of how long it takes to clear 50% of the drug after reaching Cmax. Blood samples collected pre dose and at multiple timepoints post dose will be used to determine t1/2 of belzutifan.
Steady state trough concentration (Ctrough,ss) of belzutifan after multiple doses (Cohort 1) | Pre-dose, and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours postdose
  Ctrough,ss is the lowest concentration reached by a drug before the next dose is administered. Blood samples taken at predose and at specified times post dose will be used to determine Ctrough,ss of belzutifan.
Accumulation ratio (RAC) of belzutifan after multiple doses (Cohort 1) | Pre-dose, and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours postdose
  RAC is the ratio of accumulation of a drug under steady state conditions after repeated administration as compared to a single dose. Blood samples collected pre dose and at multiple timepoints post dose will be used to determine RAC of belzutifan.
Apparent oral clearance (CL/F) of belzutifan after multiple doses (Cohort 1) | Pre-dose, and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours postdose
  CL/F is the apparent total clearance of the drug from plasma after oral administration. Blood samples collected pre dose and at multiple timepoints post dose will be used to determine CL/F of belzutifan.
Apparent oral volume (Vz/F) of belzutifan after multiple doses (Cohort 1) | Pre-dose, and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours postdose
  Vz/F is the apparent volume of distribution of the drug during terminal phase after non-intravenous administration. Blood samples collected pre dose and at multiple timepoints post dose will be used to determine Vz/F of belzutifan.

SECONDARY OUTCOMES:
Objective response rate (ORR) | Up to approximately 68 months
  ORR is defined as the percentage of participants who have a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions) per Response Evaluation Criteria In Solid Tumors 1.1 (RECIST 1.1.) The percentage of participants who experience a CR or PR as assessed by blinded independent central review based on RECIST 1.1 will be presented.
Duration of response (DOR) | Up to approximately 68 months
  For participants who demonstrate a confirmed Complete Response (CR: Disappearance of all target lesions) or confirmed Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1, DOR is defined as the time from first documented evidence of CR or PR until progressive disease (PD) or death. Per RECIST 1.1, PD was defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also have demonstrated an absolute increase of at least 5 mm. The appearance of one or more new lesions was also considered PD. The DOR as assessed by blinded independent central review will be presented.
Progression-free survival (PFS) | Up to approximately 68 months
  PFS is defined as the time from first dose of study treatment to the first documented progressive disease (PD) or death due to any cause, whichever occurs first. Per RECIST 1.1, PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions is also considered PD. PFS as assessed by blinded independent central review will be presented.
Overall survival (OS) | Up to approximately 68 months
  OS, defined as the time from first dose of study treatment to death due to any cause, will be presented.
Steady state trough concentration (Ctrough,ss) of belzutifan (Cohort 2) | Pre-dose, and 1, 2 and 4 hours postdose
  Cmin,ss is the minimum plasma drug concentration. Blood samples collected pre dose and at multiple timepoints post dose will be used to determine Cmin,ss of belzutifan.
Percent change from baseline in erythropoietin (EPO) level | Baseline, up to approximately 6 weeks
  Percent change from baseline in EPO level will be measured and presented.
Cmax,ss of belzutifan for UGT2B17 and CYP2C19 phenotypes | Week 3 Day 7: pre-dose, and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours postdose
  Cmax,ss is the maximum concentration of the drug observed in plasma. Blood samples collected pre dose and at multiple timepoints post dose will be used to determine Cmax,ss of belzutifan for participants with UGT2B17 and CYP2C19 phenotypes.
AUCss of belzutifan for UGT2B17 and CYP2C19 phenotypes | Week 3 Day 7: pre-dose, and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours postdose
  AUC0-24,ss is a measure of plasma drug concentration vs time and is estimated as the area under the plot of plasma concentration against time after drug administration. Blood samples collected pre dose and at multiple timepoints post dose will be used to determine AUC0-24,ss of belzutifan for participants with UGT2B17 and CYP2C19 phenotypes.
Ctrough,ss of belzutifan for UGT2B17 and CYP2C19 phenotypes | Week 3 Day 7: pre-dose, and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours postdose
  Ctrough,ss is the lowest concentration reached by a drug before the next dose is administered. Blood samples taken at predose and at specified times post dose will be used to determine Ctrough,ss of belzutifan for participants with UGT2B17 and CYP2C19 phenotypes.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (5):
- China (5):
  - Beijing Cancer hospital-Digestive Oncology ( Site 0001), Beijing, Beijing Municipality
  - SUN YAT-SEN UNIVERSITY CANCER CENTRE-Urology Surgery Department ( Site 0005), Guangzhou, Guangdong
  - Nanjing Drum Tower Hospital The Affiliated Hospital of Nanjing University Medical School-Urology ( S, Nanjing, Jiangsu
  - Tianjin Medical University Cancer Institute and Hospital ( Site 0003), Tianjin, Tianjin Municipality
  - The Second Affiliated hospital of Zhejiang University school of medicine-Urology ( Site 0007), Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/